CLINICAL TRIAL: NCT04520620
Title: Evaluation of the Concentration-effect Relationship of Enoxaparin for Thromboembolic Prevention in COVID-19 Intensive Unit Care Patients.
Brief Title: Concentration-effect Relationship of Enoxaparin for Thromboembolic Prevention
Acronym: COV-ENOX
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: End of the COVID 19 epidemic in the region and decision to participate in a national study on the same subject (COVI-DOSE).
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: CHU Saint-Etienne - Laboratoire de Pharmacologie - Toxicologie - Gaz du sang (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20CH089; 2020-001823-15 (EudraCT Number)
Record Dates: First submitted 2020-07-22; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-07

CONDITIONS: Sars-CoV2
Keywords: enoxaparin; intensive care unit; pharmacokinetics; SARS-Co-V-2; Lovenox
MeSH Terms: interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- enoxaparin treatment (Experimental): Patients infected by SARS-CoV-2 in intensive care unit with enoxaparin treatment will be included.
  They will have enoxaparin pharmacokinetic and ultrasound of the lower limbs at 7, 14 and 21 days after inclusion.
  Interventions: Drug: Lovenox 40 MG in 0.4 mL Prefilled Syringe; Device: Ultrasound of the lower limbs

INTERVENTIONS:
Drug: Lovenox 40 MG in 0.4 mL Prefilled Syringe — Patients with a high thrombotic risk:
  In patients with a BMI included between < 30 kg/m² and > 30 kg/m² without added thrombotic risk factor:
  * Enoxaparin 40 milligrams, (4,000 IU) twice daily subcutaneously (SC) for the entire duration of the intensive care hospitalization
  * if weight > 120 kg, enoxaparin 60 milligrams (6000 IU) twice daily subcutaneously for the entire duration of the intensive care hospitalization
  Patients with a very high thrombotic risk:
  In patients with a BMI > 30 kg/m2 with added thrombotic risk factor (active cancer, recent personal history of thromboembolic event), or if iterative or unusual catheter thromboses, or if marked inflammatory syndrome and/or hypercoagulability (e.g. fibrinogen > 8 g/L or D-Dimer > 3 μg/ml or 3000 ng/ml)
  * Enoxaparin sodium curative at a dose of 100 IU/kg/12h subcutaneously (SC) not to exceed a dose of 100 mg/12 hours
  Other Names: enoxaparin
Device: Ultrasound of the lower limbs — A 4-point compression ultrasound will be performed. In case of suspicion, an angiologist will perform to check the absence of legs thrombosis.

SUMMARY:
Patients with COVID-19 have special demographic characteristics including thromboembolic risk factors .

The pharmacokinetics of enoxaparin administered subcutaneously in the intensive care unit patient are not described.

Finally, given the lack of knowledge on the pharmacokinetic/pharmacodynamic properties of enoxaparin in intensive care unit patients infected with SARS-CoV-2, we propose to conduct a prospective multicenter cohort study to collect the biological data necessary for its study.

DETAILED DESCRIPTION:
D-dimers greater than 1 μg/mL are a prognostic factor for 28-day mortality (odds ratio=18, 2-128). The use of preventive doses of enoxaparin (4,000 to 6,000 anti-Xa per day) or unfractionated heparin (10,000 to 15,000 IU per day) has been associated with a reduction in mortality of approximately one-third in patients with D-dimer levels greater than 3 μg/mL or those with sepsis-induced coagulopathy (SIC (sepsis-induced coagulopathy) score > 4)

For the intensive care unit patient, the preventive enoxaparin dosages were increased to 4,000 anti-Xa IU twice daily and to 6,000 anti-Xa IU twice daily if the patient weighs more than 120 kg. Curative treatment is even proposed in cases of marked inflammatory syndrome and/or hypercoagulability (e.g. fibrinogen > 8 g/L or D-Dimer > 3 μg/mL or 3000 ng/mL) even without symptomatic thrombosis.

Given the lack of data on the use of these high "prophylactic" doses of enoxaparin, it is proposed that anti-Xa activity be monitored after the 3rd injection, and then regularly in the event of renal failure (because LMWHs are renally eliminated), to look for overdosage exposing a higher risk of bleeding. It is also proposed to regularly monitor (at least every 48 hours) the hemostasis of patients in search of multivisceral failure, or of coagulopathy of consumption which will require a re-evaluation of the heparin therapy dosage, these events being associated with an increased risk of haemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 ans
* SARS-CoV-2 infected intensive care unit patients
* Diagnosis of SARS-CoV-2 respiratory infection was made with a nasopharyngeal swab or a deep respiratory specimen.
* Patient receiving enoxaparin treatment as part of care or as part of a clinical trial for the prevention or treatment of thromboembolic venous disease.
* Patient affiliated or entitled to a social security scheme

Exclusion Criteria:

* Creatinine clearance according to Cockcroft and Gault <30ml/min.
* Hypersensitivity to enoxaparin sodium, heparin or its derivatives, including other low molecular weight heparins (LMWHs)
* History of immune-mediated heparin-induced thrombocytopenia (HIT) in the last 100 days or in the presence of circulating antibodies
* Active clinically significant bleeding or a condition associated with a high risk of bleeding, such as a recent hemorrhagic stroke, gastrointestinal ulcer, the presence of a malignant tumour at high risk of bleeding, recent brain, spinal or ophthalmologic surgery, known or suspected esophageal varices, arteriovenous malformations, vascular aneurysm or major intrarachidian or intracerebral vascular abnormalities.
* Spinal, epidural or locoregional anaesthesia or anaesthesia when enoxaparin sodium is used for curative treatment within the previous 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-02 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Measure of anti-Xa activity | Up to 1 month
  Measure of anti-Xa activity by chromogenic method.

SECONDARY OUTCOMES:
Analysis of hemorrhagic risk | Up to 1 month
  Hemorrhagic risk is composite of :
  * Major haemorrhage as defined by the International Society on Thrombosis and Haemostasis (ISTH) definition
  * clinically significant haemorrhage
Venous thromboembolic events | Up to 1 month
  Venous thromboembolic events is composite of:
  * symptomatic or symptomatic proximal deep vein thrombosis
  * asymptomatic or symptomatic pulmonary embolism
Analysis individual patient characteristics by the biomarker of Kidney function | Up to 1 month
  Rate of creatinine.
Analysis individual patient characteristics by the biomarker of inflammation | Up to 1 month
  Biomarker of inflammation is composite of C-reactive protein (CRP) and inflammatory cytokines.
Analysis individual patient characteristics by the biomarker of coagulation | Up to 1 month
  Biomarker of coagulation is composite of fibrinogen and D-Dimers.
Demographic characteristics | Up to 1 month
  Analysis of weight, age, sex, height, presence of a high thrombotic risk factor (history of venous thrombotics, active cancer, invasive mechanical ventilation).

CONTACTS AND LOCATIONS:
Overall Officials: Paul ZUFFEREY, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (4):
- France (4):
  - Groupement Hospitalier des portes de Province, Montélimar
  - Centre Hospitalier de Roanne, Roanne
  - CHU de Saint-Etienne, Saint-Etienne
  - Clinique Mutualiste, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No